CLINICAL TRIAL: NCT02984683
Title: Open-label Phase 2 Study Evaluating Efficacy and Safety of SAR566658 Treatment in Patients With CA6 Positive Metastatic Triple Negative Breast Cancer
Brief Title: Study Evaluating Efficacy and Safety of SAR566658 Treatment in Patients With CA6 Positive Metastatic Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued considering the limited clinical benefit combined with a higher than expected rate of known non-serious ophthalmological event.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT14884; 2016-001962-27 (EudraCT Number); U1111-1182-7044 (Other: UTN)
Record Dates: First submitted 2016-12-04; First posted 2016-12-07 (Estimated); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — SAR-566658

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR566658 90 mg/m^2 (Experimental): Participants received SAR566658 90 milligram per square meter (mg/m^2) as intravenous infusion on Day 1 and Day 8 of each 21-day treatment cycle (maximum number of cycles received was 3).
  Interventions: Drug: SAR566658 (ACT14884)
- SAR566658 120 mg/m^2 (Experimental): Participants received SAR566658 120 mg/m^2 as intravenous infusion on Day 1 and Day 8 of each 21-day treatment cycle (maximum number of cycles received was 3).
  Interventions: Drug: SAR566658 (ACT14884)

INTERVENTIONS:
Drug: SAR566658 (ACT14884) — Pharmaceutical form:Solution Route of administration: Intravenous

SUMMARY:
Primary Objective:

To evaluate the tumor Objective Response Rate (ORR), according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) of SAR566658 in participants with anti-carbonic anhydrase 6 (CA6)-positive metastatic triple negative breast cancer (TNBC). Part 1: To select the SAR566658 dose based on ORR and safety of 2 dose levels of SAR566658. Part 2: Part 2a: To demonstrate the activity of SAR566658 based on ORR in participants overexpressing CA6 (membrane intensity of 2+, 3+ in greater than or equal to (>=) 30% of tumor cells) treated at the selected dose in an expanded cohort, in addition to the participants treated in Part 1. - Part 2b: To assess the efficacy in participants with metastatic TNBC and mild CA6 expression.

Secondary Objectives:

To assess:

* Disease Control Rate (DCR), Duration of Response (DOR), Progression-Free Survival (PFS), and Time To Progression (TTP).
* The impact of ocular primary prophylaxis on the incidence of keratopathies.
* The potential immunogenicity of SAR566658.
* To evaluate the global safety profile.

DETAILED DESCRIPTION:
The duration of the study for 1 participant included a screening period of up to 21 days prior to first study drug administration, 3-week treatment cycle(s) (until 30 days after last SAR566658 administration), and a follow-up period. Each participant was treated until radiological disease progression, unacceptable toxicity, or participant's refusal of further study treatment.

ELIGIBILITY:
Inclusion criteria :

* Measurable Metastatic TNBC.
* Participants with CA6-positive disease.
* Participants received at least 1 prior chemotherapy regimen but no more than 3 for advanced/metastatic disease.
* Prior anticancer therapy must have contained anthracycline (eg, doxorubicin), if not contraindicated, and a taxane (eg, docetaxel, paclitaxel) in an adjuvant/neo-adjuvant or metastatic setting.

Exclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status >=2.
* Participant less than 18 years old.
* Pregnant or breast-feeding women.
* Participants with reproductive potential who do not agree to use accepted and effective method of contraception during the study treatment period and for 6 months following discontinuation of study drug.
* Wash out period of less than 3 weeks or 5 half-lives from previous antitumor chemotherapy, immunotherapy, or any investigational treatment.
* History of brain metastasis (other than totally resected or previously irradiated and nonprogressive/relapsed), spinal cord compression or carcinomatous meningitis, or new evidence of brain leptomeningeal disease.
* Prior treatment with eribulin as last prior therapy or prior maytansinoid treatments (DM1 or DM4 antibody-drug conjugates [ADCs]).
* Known intolerance to infused protein products including other monoclonal antibodies and ADCs.
* Poor bone marrow reserve and/or poor organ function.
* Symptomatic peripheral neuropathy Grade >=2.
* Previous history of chronic corneal diseases (even if asymptomatic) or unresolved acute nonrecurrent corneal conditions.
* Participants wearing contact lenses who are not willing to stop wearing them for the duration of the study.
* Medical conditions requiring concomitant administration of strong Cytochrome P450 3A4 (CYP3A4) inhibitors, unless it could be discontinued at least 2 weeks before 1st administration of SAR566658.
* Contraindications to the use of ophthalmic vasoconstrictor and/or corticosteroid.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Investigational Site Number 0560001, Leuven, Belgium
- Investigational Site Number 2030002, Prague, Czechia
- Italy (3):
  - Investigational Site Number 3800003, Genova
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800004, Roma
- Netherlands (2):
  - Investigational Site Number 5280001, Maastricht
  - Investigational Site Number 5280002, Rotterdam
- Spain (6):
  - Investigational Site Number 7240002, Barcelona
  - Investigational Site Number 7240005, Lleida
  - Investigational Site Number 7240001, Madrid
  - Investigational Site Number 7240006, Madrid
  - Investigational Site Number 7240003, Seville
  - Investigational Site Number 7240004, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 sites in 5 countries from 23 March 2017 to 07 September 2018.
Pre-assignment Details: A total of 23 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled in the study and included in Part 1. The study was prematurely terminated due to safety reasons, hence Part 2 was not conducted and no analysis was performed.
Period: Overall Study
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Started | 11 | 12
Completed | 0 | 0
Not Completed | 11 | 12
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression | 7 | 9

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- SAR566658 90 mg/m^2: Participants received SAR566658 90 mg/m^2 as intravenous infusion on Day 1 and Day 8 of each 21-day treatment cycle (maximum number of cycles received was 3).
- Total: Total of all reporting groups
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2 | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.73 (11.23) | 50.33 (15.30) | 53.39 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigational Medicinal Product (IMP)-Related Predefined Safety Criteria Findings
Description: Predefined safety criteria was defined as occurrence of following IMP-related treatment-emergent adverse event (TEAE) (based on National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.03): Grade greater than or equal to (>=) 3 TEAE from the System Organ Class (SOC) of eye disorders, Grade >=3 peripheral neuropathy (Preferred Term), Grade >=4 TEAE. Per NCI-CTCAE v4.03, Adverse Events (AE) were graded as follows: Grade 1: Mild; asymptomatic/mild symptoms; Grade 2: Moderate; minimal, local or non-invasive intervention indicated; Grade 3: Severe or medically significant; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; Grade 5: Death related to AE.
Time Frame: Up to Cycle 2 (each cycle of 21 days)
Population: Analysis was performed on participants evaluable for predefined safety criteria population which included participants treated in the study and had completed 2 cycles, or who experienced predefined safety criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 9 | 9
Participants
  Grade>=3 related TEAE from SOC Eye disorders | 2 | 2
  Grade>=3 related peripheral neuropathy | 0 | 0
  Grade>=4 related TEAE | 0 | 0

2. Primary Outcome: Percentage of Participants With Objective Response
Description: Objective Response in participants was defined as the participants with complete response (CR) and partial response (PR) as best response according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). As per RECIST 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline, every 6 weeks until radiological disease progression or study cut-off, whichever comes first (maximum number of cycles was 3, each cycle 21 days)
Population: Analysis was performed on all-treated population which included participants who actually received at least 1 dose or any partial dose of SAR566658.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 11 | 12
percentage of participants | 9.1 [1.0 to 31.0] | 8.3 [0.9 to 28.7]

3. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control in participants was defined as the participants with CR, PR and stable disease (SD) with a duration of at least 3 months. As per RECIST 1.1, CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 2
Population: Data for this outcome measure was not collected and analyzed due to early termination of the study.
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first radiological documentation of tumor progression or death (due to any cause), whichever comes first. As per RECIST 1.1, CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 2
Population: Data for this outcome measure was not collected and analyzed due to early termination of the study.
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval between the date of first study treatment administration and the date of documented tumor progression or death (due to any cause), whichever comes first. As per RECIST 1.1, progression was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 2
Population: Data for this outcome measure was not collected and analyzed due to early termination of the study.
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time interval between the date of first study treatment administration and the date of the first radiologically documented tumor progression. As per RECIST 1.1, progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: as for outcome 2
Population: Data for this outcome measure was not collected and analyzed due to early termination of the study.
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events (SAE)
Description: AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. TEAEs were defined as AEs that developed or worsened in grade or became serious during the on-treatment period (the time from the first treatment administration to the last treatment administration +30 days). An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.
Time Frame: Up to 30 days after last drug administration (maximum number of cycles was 3, each cycle 21 days)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 11 | 12
Participants
  Any TEAE | 11 | 12
  Any treatment emergent SAE | 1 | 6
  Any TEAE leading to treatment discontinuation | 3 | 3

8. Secondary Outcome: Number of Participants With Keratopathies (Corneal Toxicity)
Description: Keratopathy is an eye disorder that involves a blister-like swelling of the cornea (the clear layer in front of the iris and pupil). All participants received ocular primary prophylaxis in each eye in order to prevent the occurrence of keratopathies at the time of each infusion (vasoconstrictor, ophthalmic topical steroid, and cold mask on eyes) and steroid eye drops for an additional 2 days following SAR566658 administration.
Time Frame: Up to 30 days after last drug administration (maximum number of cycles was 3, each cycle 21 days)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 11 | 12
Participants | 3 | 5

9. Secondary Outcome: Number of Participants With Positive Anti-SAR566658 Antibodies Response
Time Frame: Up to 3 treatment cycles, each cycle 21 days
Population: Data for this outcome measure was not collected and analyzed due to early termination of the study.
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from the baseline up to 3 treatment cycles, each cycle 21 days.
Description: Reported AEs are TEAEs i.e. AEs that developed/worsened during 'treatment period'(time from the first treatment administration to the last treatment administration + 30 days). Analysis was performed on safety population which included all participants who received at least 1 dose (or any partial dose) of SAR566658.
Arm/Group | SAR566658 90 mg/m^2 | SAR566658 120 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/11 | 6/12
Other Adverse Events (participants affected / at risk) | 11/11 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR566658 90 mg/m^2 (N=11) | SAR566658 120 mg/m^2 (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR566658 90 mg/m^2 (N=11) | SAR566658 120 mg/m^2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear Pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1)
Abnormal Sensation In Eye (Eye disorders) | 1 (1) | 1 (1)
Corneal Epithelial Microcysts (Eye disorders) | 0 (0) | 1 (1)
Corneal Opacity (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 3 (3) | 1 (1)
Halo Vision (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 5 (5) | 1 (1)
Keratopathy (Eye disorders) | 3 (3) | 5 (6)
Periorbital Oedema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 1 (1)
Vitreous Floaters (Eye disorders) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 3 (3)
Device Related Thrombosis (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 2 (2) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2)
Neuropathy Peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued considering the limited clinical benefit combined with higher than expected rate of known non-serious ophthalmological event, hence Part 2 was not conducted and some of pre-specified endpoints were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02984683/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT02984683/SAP_001.pdf